CLINICAL TRIAL: NCT00801957
Title: A Double Blind, Multicentre, Randomised, Parallel Group Study to Demonstrate the Equivalence of the Response to Vaccination of a Tacrolimus Ointment Regimen to a Steroid Ointment Regimen in Children With Moderate to Severe Atopic Dermatitis
Brief Title: Equivalence of the Response to Vaccination of Tacrolimus Ointment to a Steroid Ointment Regimen in Children With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FG-506-06-27
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; meningitis; vaccination; tacrolimus; steroids; equivalence response; meningococcal vaccine
MeSH Terms: conditions — Dermatitis, Atopic; Meningitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): tacrolimus ointment 0.03%
  Interventions: Drug: tacrolimus ointment 0.03%; Biological: Meningitec; Biological: AC VAX
- 2 (Active Comparator): hydrocortisone acetate 1% and butyrate 0.1%
  Interventions: Drug: hydrocortisone acetate ointment 1%; Drug: hydrocortisone butyrate ointment 0.1%; Biological: Meningitec; Biological: AC VAX
- 3 (Other): Control group vaccination and challenge dose only
  Interventions: Biological: Meningitec; Biological: AC VAX

INTERVENTIONS:
Drug: tacrolimus ointment 0.03% — topical application
  Other Names: Protopic 0.03%
  Arms: 1
Drug: hydrocortisone acetate ointment 1% — topical application
  Other Names: ATC code H02AB09
  Arms: 2
Drug: hydrocortisone butyrate ointment 0.1% — topical application
  Other Names: ATC code H02AB09
  Arms: 2
Biological: Meningitec — im injection
Biological: AC VAX — im injection

SUMMARY:
Seven-month study in pediatric patients (2-11 years) with moderate to severe AD who were considered to benefit from vaccination to prevent invasive disease caused by Neisseria meningitides serogroup C.

DETAILED DESCRIPTION:
At the week 1 visit, the patients were vaccinated with a protein-conjugated vaccine against meningitis. All patients received a challenge at the month 6 visit with a low dose of meningo polysaccharide vaccine. A control group of healthy subjects (not suffering from atopic dermatitis) received only the vaccination and the challenge dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe atopic dermatitis and in need for treatment
* Patients require vaccination to prevent invasive disease caused by Neisseria meningitidis serogroup C

Exclusion Criteria:

* Patients have known hypersensitivity to macrolides, tacrolimus and any component of the vaccine
* Patients have an acute severe febrile illness, genetic epidermal barrier defect such as Netherton's syndrome or generalized erythroderma, a skin infection on the affected and to be treated area
* Patients have already received a meningo polysaccharide or conjugated vaccine against meningitis

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2003-03; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with serum bactericidal antibody titer of ≥ 8 | 5 weeks

SECONDARY OUTCOMES:
Assessment of other immunological parameters | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (33):
- Australia (9):
  - Kogarah, New South Wales
  - St Leonards, New South Wales
  - Benowa, Queensland
  - Carina Heights, Queensland
  - Herston, Queensland
  - North Adelaide, South Australia
  - Carlton, Victoria
  - Parkville, Victoria
  - Fremantle, Western Australia
- Leuven, Belgium
- Germany (5):
  - Bretten
  - Ettenheim
  - Gersfeld
  - Kehl
  - Tettnang
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
- Kopavogur, Iceland
- Saint Julians, Malta
- Poland (10):
  - Karpacz
  - Krakow
  - Lodz
  - Opole
  - Poznan
  - Rabka-Zdrój
  - Warsaw
  - Wroclaw
  - Zabrze
  - Zgierz
- Portugal (2):
  - Lisbon
  - Porto

REFERENCES:
- [Background] Hofman T, Cranswick N, Kuna P, Boznanski A, Latos T, Gold M, Murrell DF, Gebauer K, Behre U, Machura E, Olafsson J, Szalai Z; International Tacrolimus Ointment Study Group. Tacrolimus ointment does not affect the immediate response to vaccination, the generation of immune memory, or humoral and cell-mediated immunity in children. Arch Dis Child. 2006 Nov;91(11):905-10. doi: 10.1136/adc.2006.094276. Epub 2006 Jun 23. PMID 16798785